CLINICAL TRIAL: NCT06456632
Title: The Effect of Su Jok Therapy on Postoperative Pain, Anxiety and Patient Satisfaction in Benign Prostatic Hyperplasia (BPH) Patients With Transurethral Prostate Resection (TUR-P): A Randomized Controlled Study
Brief Title: The Effect of Su Jok Therapy on Postoperative Pain, Anxiety and Patient Satisfaction in Patients With BPH
Acronym: SuJokTherapy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KA24/89; KA24/89 (Other Grant/Funding Number: Baskent University Institutional Ethics Committee)
Record Dates: First submitted 2024-05-30; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Transurethral Resection (TUR) Syndrome
Keywords: Su jok therapy; Pain; Anxiety; Patient Satisfaction; Nursing
MeSH Terms: conditions — Syndrome; Pain; Anxiety Disorders; Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: Intervention and Control group
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Group not receiving Su Jok Therapy
- Intervention Group (Experimental): Group receiving Su jok therapy
  Interventions: Other: Intervention Su Jok Therapy

INTERVENTIONS:
Other: Intervention Su Jok Therapy — Su Jok Therapy
  Arms: Intervention Group

SUMMARY:
This study is the first nursing study in the field of urology to examine the effect of Su Jok Therapy on postoperative pain, anxiety and patient satisfaction in patients who underwent Transurethral Resection of the Prostate with a diagnosis of BPH and is thought to make an important contribution to evidence-based nursing practices. In line with the results obtained from the study, it is expected that the anxiety levels of patients planned to apply Su Jok therapy will be reduced, pain levels will be reduced, and patient satisfaction will increase.

DETAILED DESCRIPTION:
Considering the literature, it is seen that the number of studies examining the effects of integrative methods used in symptom management such as Su Jok Therapy on postoperative pain, anxiety and patient satisfaction are high and have positive effects as a result. Still, there are a limited number of studies on the effects of Su Jok Therapy on postoperative pain and anxiety in the surgical field. This study is thought to make an important contribution to evidence-based nursing practices as it is the first nursing study in the field of urology to examine the effect of Su Jok Therapy on postoperative pain, anxiety level and patient satisfaction in patients undergoing transurethral resection of the prostate (TUR-P) with a diagnosis of BPH. In line with the results obtained from the study, it is planned to reduce the anxiety and pain levels of patients who are planned to apply Su Jok therapy and to increase patient satisfaction. In this study, it is aimed to determine the effect of Su Jok Therapy on postoperative pain, anxiety and patient satisfaction in patients diagnosed with BPH who underwent Transurethral Resection of Prostate (TUR-P).

Research Hypotheses:

H0-1: Su Jok therapy is not effective in reducing postoperative pain level in patients undergoing TUR-P.

H1-1: Su Jok therapy is effective in reducing postoperative pain level in patients undergoing TUR-P.

H0-2: Su Jok therapy is not effective in reducing anxiety level in patients undergoing TUR-P.

H1-2: Su Jok therapy is effective in reducing anxiety level in patients undergoing TUR-P.

H0-3: Su Jok therapy is not effective in increasing patient satisfaction in patients undergoing TUR-P.

H1-3: Su Jok therapy is effective in increasing patient satisfaction in patients undergoing TUR-P.

The population of this study will consist of patients who applied to the Urology Outpatient Clinic of Başkent University Ankara Hospital and were planned to undergo Transurethral Prostate Resection for the first time with the diagnosis of BPH.

According to hospital records, 52 patients diagnosed with BPH underwent TUR-P in the last year. The sample size of the study was calculated by a statistical expert using a sample size calculation program (G*Power version 3.1.9.4). The minimum sample size required for the study was planned to include at least 52 patients (26 intervention, 26 control) to be approximately equally distributed in the groups that will provide 80% test power at 95% confidence level, with an effect size of 0.80 and Cohen's large effect size of 0.80 for "One-Way Analysis of Variance" when the parametric test assumptions of "Whether there is a difference between more than two groups" are met, and "Kruskal Wallis Test" when not met.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older diagnosed with BPH,
* First time undergoing TUR-P surgery,
* Does not have any cognitive, affective and verbal communication problems that prevent understanding of the information given and expressing the pain and anxiety correctly,
* Patients who volunteered to participate in the study

Exclusion Criteria:

* Those who have loss of sensation, amputation, injury, wound, active burn, fungal disease, etc. in their hands that will prevent them from practicing,
* HbA1c value in patients diagnosed with diabetes mellitus: 6.5% and above
* Using any complementary and integrative health practice in the last 3 months,
* Patients who do not speak Turkish, have hearing problems, language problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Patient Pain Assessment | From preoperative to 8 hours postoperatively
  Patient's pain will be assessed. The Visual Analogue Scale (VAS) will be used to assess pain.The Visual Analogue Scale (VAS) measures pain intensity. The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be'). Ask the patient to rate their current level of pain by placing a mark on the line.
Anxiety | Preoperative and 8th hour after surgery
  Patient's anxiety will be assessed. The State Anxiety Inventory (SAI) will be used to assess anxiety. The State Anxiety Inventory (SAI) is a commonly used measure of trait and state anxiety. It can be used in clinical settings to diagnose anxiety and to distinguish it from depressive syndromes. It also is often used in research as an indicator of caregiver distress. its most popular version, has 20 items for assessing trait anxiety and 20 for state anxiety.
Patient satisfaction | 8th hour after surgery
  Patient satisfaction will be assessed. Visual Analog Patient Satisfaction Scale will be used to evaluate patient satisfaction.This scale ranges from 0 (not satisfied at all) to 10 (very satisfied).